CLINICAL TRIAL: NCT02026284
Title: Factors Affecting Anesthesia Preferences of Gravid Women Who Are to Deliver by Caesarean Section
Brief Title: Factors Affecting Anesthesia Preferences of Gravid Women
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Sanem Cakar Turhan, Specialist, Ankara University
Other Study IDs: 38-828
Record Dates: First submitted 2013-12-27; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Caesarean Section, Anaesthesia, Questionnaires
Keywords: Caesarean section; Anaesthesia; Questionnaires
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gravid women: A questionnaire was performed to gravid women
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire was performed to gravid women who are to deliver, regarding theri anesthesia preferences.

SUMMARY:
The investigators aim to evaluate the preferences for anaesthesia methods of gravid women who are to deliver baby by caesarean section, the rates of general anaesthesia and regional anaesthesia, the reasons for preferences of general anaesthesia and regional anaesthesia and the factors affecting these preferences.

A questionnaire consisting of 20 questions were applied to gravid women applying for delivery by elective caesarean operation, at Ankara University Faculty of Medicine Hospital for Gynaecology and Obstetrics between February 2010 and February 2011, in order to study the anaesthesia technique the patients prefer and the reason behind their preferences. Those gravid women who accepted to take part in the study were provided information about the questionnaire and their oral and written approvals were obtained.

DETAILED DESCRIPTION:
The questionnaire was applied to the patients in visit queue a day before or while the patients were in waiting room for caesarean operation. The gravid women who were between 26th and 40th week of their pregnancy were included in the questionnaire. Those who were taken into emergency service, those with communication problems, those whose mental conditions deter them to answer questions and those who did not want to answer the questions on the questionnaire were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* gravid women who were between 26th and 40th week of their pregnancy were included in the questionnaire.

Exclusion Criteria:

* gravid women who were taken into emergency service, those with communication problems, those whose mental conditions deter them to answer questions and those who did not want to answer the questions on the questionnaire

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A questionnaire consisting of 20 questions were applied to gravid women applying for delivery by elective caesarean operation, at Ankara University Faculty of Medicine Hospital for Gynaecology and Obstetrics between February 2010 and February 2011
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who prefer regional anesthesia and who prefer general anesthesia | 1 day

SECONDARY OUTCOMES:
Factors affecting the preference of regional anesthesia and general anesthesia | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Helin Sahintürk, Specialist, Principal Investigator — Ankara University Medical School Anesthesiology and ICU
Locations (1):
- Ankara University Medical School Anesthesiology and ICU Department, Ankara, Turkey (Türkiye)